CLINICAL TRIAL: NCT05641649
Title: Bioequivalence Study of Sodium Valproate and Valproic Acid Extended Release Tablets in Healthy Human Volunteers
Brief Title: Bioequivalence Study of Sodium Valproate and Valproic Acid Tablets
Acronym: BA-BE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kathmandu University (Other)
Collaborators: Asian Pharmaceuticals Pvt. Ltd. (Industry)
Responsible Party: Principal Investigator, Rajani Shakya, Associate Professor, Kathmandu University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BE-001-022
Record Dates: First submitted 2022-11-10; First posted 2022-12-08 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Epilepsy
Keywords: Bioequivalence; Pharmacokinetics; Valproic acid; Sodium valproate
MeSH Terms: conditions — Epilepsy | interventions — Valproic Acid

STUDY DESIGN:
Intervention Model Description: On the first study day, volunteers will be grouped into two. One group will be given test formulation and other will be given innovator formulation. Simple randomization technique will be used for this. Predose blood sample will be collected 15 minutes before drug administration. Later 3 ml blood sample will be collected at 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 60 and 72 hours after drug administration.
  After giving a washout period of 7 days, group of volunteers who have received test formulation on first study day will be given innovator and those who received innovator on the first study day will be given test formulation on the second study day.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test formulation group of volunteers (Experimental): Sixteen healthy subjects aged between 18 and 60 years who satisfy the inclusion/ exclusion criteria will be enrolled in the study. Volunteers will be assigned to take particular formulation by a method of randomization on the first study day.
  Half of the volunteers falling in the test formulation arm will be given a tablet of test formulation with 200 ml of water in an empty stomach on the first study day. In the second study day, these volunteers will be exchanging the formulations.
  Interventions: Drug: Sodium valproate and valproic acid extended release tablet
- Innovator formulation group of volunteers (Experimental): Sixteen healthy subjects aged between 18 and 60 years who satisfy the inclusion/ exclusion criteria will be enrolled. Volunteers will be assigned to take particular formulation by a method of randomization on the first study day.
  Half of the volunteers falling in the innovator formulation arm will be given a tablet of innovator formulation with 200 ml of water in an empty stomach on the first study day. In the second study day, these volunteers will be exchanging the formulations.
  Interventions: Drug: Sodium valproate and valproic acid extended release tablet

INTERVENTIONS:
Drug: Sodium valproate and valproic acid extended release tablet — Test or innovator tablet formulation of sodium valproate and valproic acid will be administered orally to the volunteers on each study days in fasting condition. Volunteers will be receiving a single tablet of either of the formulations on the study days by a randomization technique so that each of them receives both formulations during the study period.
  Other Names: Test drug: VALPROT 500XR; Reference drug: Encorate chrono 500

SUMMARY:
Bioavailability is the extent and rate to which the active drug ingredient or active moiety from the drug product is absorbed and becomes available at the site of drug action. Bioavailability of an active substance delivered from a pharmaceutical product should be known and reproducible. In the past, several therapeutic misadventures related to differences in bioavailability affirm to the necessity of testing the performance of dosage forms in delivering the active substance to the systemic circulation and thereby to the site of action. If there is no clinically significant difference in the bioavailability of two medicines they are considered to be bioequivalent.

The bioavailability and bioequivalence studies of various drug candidates have been routine regulatory requirements in many countries for licensing of the drug product. Department of Drug Administration, Ministry of health and Population has encouraged Nepalese Pharmaceutical Industries legally to submit pharmacokinetic data where possible for licensing purpose for certain drug candidates and their dosage forms. The comparative in-vivo bioequivalence study is necessary for those products which have low therapeutic index, low bioavailability, non-linear kinetics, poor dissolution profile, variable bioavailability and/or bioequivalence. Department of Drug Administration necessitated bioequivalence and bioavailability study for the modified release dosage form of those drug molecules whose blood steady state concentration is of great importance, e.g. sodium valproate, valproic acid, carbamazepine, antibiotics etc. Considering the need to confirm safety and effectiveness of the medications and also for the regulatory requirement, this study to assess the bioequivalence of sodium valproate and valproic acid extended release tablet manufactured by a Nepalese pharmaceutical company, Asian Pharmaceuticals Pvt. Ltd., with an innovator formulation is being carried out in healthy human volunteers.

DETAILED DESCRIPTION:
Successful therapeutic management of patients with epilepsy requires selection of an appropriate antiepileptic regimen, optimal dosing and patient compliance. Valproate is primarily used to treat epilepsy and bipolar disorder. Valproate exists in two main molecular variants; sodium valproate and valproic acid. These molecules have been widely used in the last decade and is now considered as relatively safe and effective anticonvulsant agents. These drug molecules were registered in Department of Drug administration of Nepal long time back.

The mechanism of action of valproate is not clear. There are three proposed mechanism of action: 1) It increases the brain γ-aminobutyric acid (GABA), 2) It potentiates the postsynaptic response to GABA, and 3) It exerts a direct membrane effect.

Valproate can be administrated by intravenous, oral and rectal routes. Among them, the oral route is mostly and widely used. Valproate is highly bound (90%) to human plasma albumin at therapeutic concentrations. This property tends to keep most of the drug within the vascular compartment. The clearance of valproate is independent of liver blood flow but is highly dependent on the free fraction. It has been recognized that the blood levels-dose relationship for valproate is highly variable among patients. Valproate is eliminated almost exclusively by hepatic metabolism (>96% of administered dose).

Sodium valproate and valproic acid are the critical dose medicines. Critical dose medicines are those medicines for which relatively small variations in plasma concentrations may cause significant adverse effects or loss of efficacy. Stable serum levels of valproic acid without marked peak-to-trough fluctuations, reduced frequency of dosing, and the possibility of dosing flexibility will improve cure rate, patient compliance, satisfaction and, ultimately, quality of life. Valproic acid is available in different dosage forms for parenteral and oral use. All available oral formulations are almost completely bioavailable, but they differ in dissolution characteristics and absorption rates. Extended-release formulations can be very helpful in achieving above mentioned objectives and avoiding consequences due to differences in dissolution characteristics.

"VALPROT 500XR" is the extended release formulation of sodium valproate and valproic acid manufactured in Nepal by Asian Pharmaceuticals Pvt. Ltd. Due to presence of several brands of these molecules in the market, there is possibility of brand substitution in patients. If the newer brand has different pharmacokinetic property and bioavailability than the conventional ones then this can lead to several problems like loss of seizure control, seizure related injury, accidents etc. So, it is prudent to ensure that the values for pharmacokinetic parameters of existing formulations and the newly designed formulation are comparable with each other. Yet there is no information available on pharmacokinetic profile of this new extended release formulation. Therefore, there is a strong need of a bioequivalence study to make comparison of pharmacokinetic profile of "VALPROT 500XR" and the marketed innovator brand to prove them interchangeable.

Bioequivalence means the absence of greater-than-allowable difference between the systemic bioavailability of a test product and that of an innovator product. The United States Food and Drug Administration (US FDA) has defined bioequivalence as 'the absence of a significant difference in the rate and extent to which the active ingredient or active moiety in pharmaceutical equivalents or pharmaceutical alternatives becomes available at the site of drug action when administered at the same molar dose under similar conditions in an appropriately designed study'. The FDA considers two products bioequivalent if the 90% confidence interval of the relative mean plasma concentration (Cmax), area under the serum drug concentration versus time curve from zero time to 24 hours (AUC0-24) and area under the serum drug concentration versus time curve from zero time to infinity (AUC0-∞) of the test to innovator product is within 80% to 125%. For narrow therapeutic index drugs where small differences in dose or blood concentration may lead to serious therapeutic failures and/or adverse drug reactions, this difference in blood concentrations or drug exposure might not be unacceptable and a narrow limit for bioequivalence is proposed.

Bioequivalence is the important tool to characterize the therapeutic efficacy of the drug product. The objective of the bioequivalence study is to provide assurance of switchability between various formulations in the interest of clinical safety. Switchability actually demands that, within the same patient, the drug concentration of the test formulation remain within the same therapeutic window achieved by the innovator formulation.

The main objective of this study is to investigate the bioequivalence of sodium valproate and valproic acid extended release tablets (VALPROT 500XR), manufactured by Asian Pharmaceuticals Pvt. Ltd. with an innovation brand having the same composition, following a single, oral dose administered.

This is an open-label, randomized, two-way crossover study comprising sixteen healthy volunteers between 18 and 60 years of age. Potential subjects will be recruited via local advertisement. Dropouts will be replaced if the number of evaluable subjects drops below 16.

Subjects meeting set inclusion criteria will be enrolled in the study after obtaining informed written consent. Complete physical examination will be carried out at the time of initial screening and also within 24 hours after each dose whenever required. Laboratory tests including liver function and renal function tests will be carried out at the time of initial screening, prior to the administration of each dose. If any person has abnormal liver function (abnormal level of liver enzymes) and/or abnormal renal function (abnormal creatinine and urea level), he/she will be withdrawn from the study.

On the first study day, volunteers will be grouped randomly into two groups. One group will be given test formulation and other will be given reference formulation. Exactly 15 minutes before the first dose, 3 ml blood sample will be collected and later at 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 60 and 72 hours after drug administration.

After giving a washout period of 7 days, on the second study day, volunteers will exchange the formulations.

Blood sample will be collected in vacutainer tubes with no anticoagulant. It will be allowed to clot at room temperature for 20 minutes. Then blood sample will be centrifuged at 3000 rpm for 15 minutes. Serum will be transferred into a separate serum container and will be promptly frozen at -20 degree Celsius until assay. Plasma samples will be analyzed using a validated bioanalytical method in the analytical laboratory of Kathmandu University. The single-dose pharmacokinetic parameters that will be evaluated include Cmax, AUC0-24, AUC0-∞, and the elimination half-life (t1/2).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 - 60 years.
2. Gender: Male / female or both
3. Weight: At least 50 kg (110 lbs) and within 15% of Ideal Body Weight (IBW). BMI between 18.0 and 29.9 kg/m², inclusive
4. All subjects should be judged normal and healthy during a pre-study medical evaluation (physical examination, including vital signs, laboratory evaluations, 12-lead ECG, hepatitis B, hepatitis C and HIV tests) performed within 14 days of the initial dose of study medication.
5. Consent: Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent (signed and dated) obtained

Exclusion Criteria:

1. Social Habits:

   i. Use of any tobacco products within month of the start of the study. ii. Ingestion of any alcoholic, caffeine- or xanthine-containing food or beverage within 48 hours prior to the initial dose of study medication.

   iii. Ingestion of any vitamins or herbal products within 7 days prior to the initial dose of the study medication.

   iv. Any recent, significant change in dietary or exercise habits. v. History of drug and/or alcohol abuse.
2. Medications:

   i. Use of any prescription or over-the-counter (OTC) medications within 14 days prior to the initial dose of study medication.

   ii. Use of any medication known to alter hepatic enzyme activity within 28 days prior to the initial dose of study medication.
3. Diseases:

   i. History of any significant cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic disease.

   ii. Acute illness at the time of either the pre-study medical evaluation or dosing.

   iii. A positive HIV, hepatitis B, or hepatitis C tests.
4. Abnormal and clinically significant laboratory test results:

   i. Clinically significant deviation from the Guide to Clinically Relevant Abnormalities.

   ii. Abnormal and clinically relevant ECG tracing.
5. Clinical Studies i. Participation in any clinical study (inclusive of final post-study examination) within the 12 weeks before screening visit.

   ii. Subject whose participation in this study will result in a participation in more than four studies over a twelve month period.
6. Donation or loss of a significant volume of blood or plasma (> 450 mL) within 28 days prior to the initial dose of study medication.
7. Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.
8. Allergy or hypersensitivity to valproic acid / sodium valproate or any other related products.
9. History of difficulties in swallowing, or any gastrointestinal disease which could affect the drug absorption.
10. Consumption of grapefruit or grapefruit containing products within 7 days of drug administration.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-08-06 (Actual); Primary Completion 2023-10-13 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Collected blood samples will be analyzed using a validated bioanalytical method to investigate bioequivalence of test and innovator formulations. If the formulations are found to be bioequivalent these will be considered interchangeable in clinical use. | Blood samples will be collected for up to 24 hours of administration of formulations in both study days. Blood sample analysis, determination of pharmacokinetic parameters and statistical analysis to evaluate bioequivalence will take nearly 2 months.
  For determining bioequivalence of test and innovator formulations, serum drug concentration will be estimated initially. Using this data, other pharmacokinetic parameters will also be estimated like time to peak concentration (tmax), elimination half-life (T1/2), area under the serum drug concentration versus time curve from zero time to 24 hrs (AUC(0-24)), area under the plasma concentration-time curve from zero to infinity (AUC 0-∞), and the elimination half-life (t1/2), using a standard pharmacokinetic software.
  Test and innovator formulation will be considered bioequivalent if the 90% confidence interval of the ratio of a log-transformed exposure measure (AUC and/or Cmax) falls within the range 80-125%.

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) | Blood samples collection up to 24 hours of drug administration
  The highest concentration of a drug in the blood after administration of test and innovator formulations
Area under the plasma concentration-time curve from zero to infinity (AUC 0-∞) | Blood samples collection up to 24 hours of drug administration
  Actual body exposure to drug after administration of test and innovator formulations in infinite time
Area under the plasma concentration-time curve from zero to 24 hours (AUC 0-24) | Blood samples collection up to 24 hours of drug administration
  Actual body exposure to drug after administration of test and innovator formulations in 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rajani Shakya, PhD, Principal Investigator — Kathmandu University
Locations (2):
- Nepal (2):
  - Department of Pharmacy, Kathmandu University, Dhulikhel, Bagmati
  - Dhulikhel Hospital, Kathmandu University Teaching Hospital, Dhulikhel, Bagmati

IPD SHARING:
Plan to Share IPD: No
The report of this study will be submitted to the sponsor company who will be further submitting to the Department of Drug Administration, the drug regulatory body in Nepal.
  The result of this study will be disseminated later in the form of research papers.

REFERENCES:
- [Background] Bialer M. Extended-release formulations for the treatment of epilepsy. CNS Drugs. 2007;21(9):765-74. doi: 10.2165/00023210-200721090-00005. PMID 17696575
- [Background] Perucca E. Extended-release formulations of antiepileptic drugs: rationale and comparative value. Epilepsy Curr. 2009 Nov-Dec;9(6):153-7. doi: 10.1111/j.1535-7511.2009.01326.x. PMID 19936129
- [Result] Dutta S, Reed RC, Cavanaugh JH. Absolute bioavailability and absorption characteristics of divalproex sodium extended-release tablets in healthy volunteers. J Clin Pharmacol. 2004 Jul;44(7):737-42. doi: 10.1177/0091270004266782. PMID 15199078
- [Result] Fujii A, Yasui-Furukori N, Nakagami T, Niioka T, Saito M, Sato Y, Kaneko S. Comparative in vivo bioequivalence and in vitro dissolution of two valproic acid sustained-release formulations. Drug Des Devel Ther. 2009 Feb 6;2:139-44. doi: 10.2147/dddt.s3556. PMID 19920901
- [Result] Yasui-Furukori N, Saito M, Nakagami T, Niioka T, Sato Y, Fujii A, Kaneko S. Different serum concentrations of steady-state valproic acid in two sustained-release formulations. Psychiatry Clin Neurosci. 2007 Jun;61(3):308-12. doi: 10.1111/j.1440-1819.2007.01656.x. PMID 17472600
- [Result] Dulac O, Alvarez JC. Bioequivalence of a new sustained-release formulation of sodium valproate, valproate modified-release granules, compared with existing sustained-release formulations after once- or twice-daily administration. Pharmacotherapy. 2005 Jan;25(1):35-41. doi: 10.1592/phco.25.1.35.55626. PMID 15767218
- [Result] Roberts D, Easter D, O'Bryan-Tear G. Epilim chrono: a multidose, crossover comparison of two formulations of valproate in healthy volunteers. Biopharm Drug Dispos. 1996 Mar;17(2):175-82. doi: 10.1002/(SICI)1099-081X(199603)17:23.0.CO;2-J. PMID 8907724